CLINICAL TRIAL: NCT03302416
Title: In Vivo Imaging of Corticotropin-releasing Factor - Nociceptin Receptor Interactions
Brief Title: CRF - Nociceptin Receptor Interactions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rajesh Narendran, Visiting Professor in Radiology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO16030242; R21DA042633 (NIH)
Record Dates: First submitted 2017-09-29; First posted 2017-10-05 (Actual); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Healthy
MeSH Terms: interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Baseline [C-11]NOP-1A scan Post-hydrocortisone [C-11]NOP-1A scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [C-11]NOP-1A PET Scan conditions (Experimental): Baseline condition and Post-hydrocortisone (1 mg/Kg, intravenous) condition
  Interventions: Drug: Hydrocortisone; Radiation: [C-11]NOP-1A

INTERVENTIONS:
Drug: Hydrocortisone
Radiation: [C-11]NOP-1A

SUMMARY:
To determine if [C-11]NOP-1A receptor binding (VT) can be altered by an intravenous hydrocortisone (cortisol) challenge through CRF-NOP interactions

DETAILED DESCRIPTION:
Examines changes in [C-11]NOP-1A pharmacokinetics caused by an intravenous hydrocortisone challenge (1 mg/kg)

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 40 years old

Exclusion Criteria:

* Current DSM-5 psychiatric disorders
* Binge drinking as defined in NIAAA criteria in the past month
* Recreational abuse of opiates, sedative-hypnotics, cocaine, amphetamines, MDMA, and PCP, as well as cannabis use
* Currently on any prescription medical or psychotropic medication;
* Current or past severe medical, endocrine, cardiovascular, immunological or neurological illnesses
* Currently pregnant or breast-feeding;
* History of radioactivity exposure via prior nuclear medicine studies or occupational exposure in past twelve months
* Metallic objects in the body that are contraindicated for MRI;
* First-degree relative with psychosis or mood disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flanigan M, Tollefson S, Himes ML, Jordan R, Roach K, Stoughton C, Lopresti B, Mason NS, Ciccocioppo R, Narendran R. Acute Elevations in Cortisol Increase the In Vivo Binding of [11C]NOP-1A to Nociceptin Receptors: A Novel Imaging Paradigm to Study the Interaction Between Stress- and Antistress-Regulating Neuropeptides. Biol Psychiatry. 2020 Mar 15;87(6):570-576. doi: 10.1016/j.biopsych.2019.09.013. Epub 2019 Sep 25. PMID 31706582

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 subjects screened, 19 assigned to interventions
Groups:
- [C-11]NOP-1A PET Scan Conditions: Baseline condition and Post-hydrocortisone (1 mg/Kg, intravenous) condition
  Hydrocortisone
  [C-11]NOP-1A
Period: Overall Study
Arm/Group | [C-11]NOP-1A PET Scan Conditions
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | [C-11]NOP-1A PET Scan Conditions
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Weight [Mean (Standard Deviation); unit: Kilograms] | 77 (16)

OUTCOME MEASURES:

1. Primary Outcome: [C-11]NOP-1A Volume of Distribution Expressed Relative to Total Plasma Concentration
Description: VT is the volume of distribution expressed relative to total plasma concentration. This is defined consistent with that reported in Consensus nomenclature for in vivo imaging of reversibly binding radioligands (Reference: J Cereb Blood Flow Metab 2007 Sep;27(9):1533-9. doi: 10.1038/sj.jcbfm.9600493)
Time Frame: Baseline and 3.5 hours post-hydrocortisone
Measure: Mean (Standard Deviation); unit: mL/cm^3
Groups:
- Baseline Participants: Healthy Controls
Arm/Group | Baseline Participants
Number analyzed (Participants) | 19
mL/cm^3
  Amygdala/baseline | 16.3 (1.9)
  Amygdala/post-hydrocortisone | 18.7 (2.8)
  Hippocampus/baseline | 11.6 (1.3)
  Hippocampus/post-hydrocortisone | 13.3 (2.0)
  Midbrain/baseline | 9.4 (1.0)
  Midbrain/post-hydrocortisone | 10.6 (1.6)
  Vental striatum/baseline | 15.1 (1.7)
  Ventral striatum/post-hydrocortisone | 17.1 (2.1)
  Caudate/baseline | 12.7 (1.4)
  Caudate/post-hydrocortisone | 14.0 (1.9)
  Putamen/baseline | 14.3 (1.6)
  Putamen/post-hydrocortisone | 16.0 (2.0)
  dorsolateralPFC/baseline | 14.4 (1.8)
  dorsolateralPFC/post-hydrocortisone | 16.4 (2.4)
  Orbital frontal cortex/baseline | 14.9 (1.8)
  Orbital frontal cortex/post-hydrocortisone | 17.1 (2.6)
  MedialPFC/baseline | 14.3 (1.8)
  MedialPFC/post-hydrocortisone | 16.2 (2.4)
  anterior cigulate/baseline | 14.6 (1.7)
  anterior cingulate/post-hydrocortisone | 16.6 (2.6)
  Cerebellum/baseline | 8.2 (0.9)
  Cerebellum/post-hydrocortisone | 9.3 (1.3)
Statistical Analysis 1: Comparison: Baseline Participants; Test type: Superiority — Baseline scan VT vs. Post-hydrocortisone scan VT; p = 0.005, Linear mixed model

ADVERSE EVENTS:
Time Frame: < 7 days
Arm/Group | [C-11]NOP-1A PET Scan Conditions
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT03302416/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT03302416/ICF_001.pdf